CLINICAL TRIAL: NCT03951402
Title: Investigation of the Effect on the QT/QTc Interval After Multiple Dose Oral Administration (100 and 200 mg Bid) of CG5503 PR in a Randomised, Double-blind, Double-dummy Placebo- and Moxifloxacin-controlled 4- Way Cross-over Phase I Study in 48 Healthy Male and Female Volunteers
Brief Title: Effect of a Multiple-dose Oral Administration of CG5503 PR on the Electrical Activity of the Heart in 48 Healthy Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HP5503/10; PK614 (Other: Sponsor code)
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Prolonged QTc Interval; Pharmacokinetic
Keywords: QT/QTc Interval
MeSH Terms: interventions — Tapentadol; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This study was a randomized, double-blind, double-dummy, placebo- and moxifloxacin-controlled, 4-way cross-over study. The randomization was in the ratio 1:1:1:1. In all treatments the amount of administered tablets and capsules were the same. At the lower dose step the amount of tablets/capsules was adjusted with matching placebos. All study procedures were the same, irrespective of whether active compound, positive control or placebo was administered.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CG5503 PR 100 mg twice daily (tapentadol hydrochloride) (Experimental): Each participant received a morning and an evening dose of 100 mg CG5503 PR on days 1 and 2 and a morning dose on Day 3 (each dose: 1 tablet CG5503 PR and 1 placebo-tablet, matching CG5503 PR); additionally at each dosing each participant received 2 placebo-capsules, matching moxifloxacin 400 mg.
  The participants received 2 tablets and 2 capsules at each dosing with approximately 150 ml water.
  Interventions: Drug: 100 mg CG5503 (tapentadol hydrochloride) PR tablet; Drug: Placebo matching CG5503 PR tablet; Drug: Placebo matching moxifloxacin capsule
- CG5503 PR 200 mg twice daily (tapentadol hydrochloride) (Experimental): Each participant received a morning and an evening dose of 200 mg CG5503 PR on days 1 and 2 and a morning dose on Day 3 (each dose: 2 tablets CG5503 PR); additionally at each dosing each participant received 2 placebo-capsules, matching moxifloxacin.
  The participants received 2 tablets and 2 capsules at each dosing with approximately 150 ml water.
  Interventions: Drug: 100 mg CG5503 (tapentadol hydrochloride) PR tablet; Drug: Placebo matching moxifloxacin capsule
- Placebo (Placebo Comparator): Each participant received a morning and an evening dose of placebo to CG5503 PR on days 1 and 2 and a morning dose on Day 3 (each dose: 2 tablets placebo, matching CG5503 PR); additionally at each dosing each participant received 2 placebo-capsules, matching moxifloxacin.
  The participants received 2 tablets and 2 capsules at each dosing with approximately 150 ml water.
  Interventions: Drug: Placebo matching CG5503 PR tablet; Drug: Placebo matching moxifloxacin capsule
- Moxifloxacin 800 mg single dose (Active Comparator): Each participant received a morning and an evening dose of placebo to CG5503 PR on days 1 and 2 and a morning dose on Day 3 (each dose: 2 tablets placebo, matching CG5503 PR); and 2 placebo-capsules, matching moxifloxacin on days 1 and 2; In the morning of Day 3, each participant received additionally 2 capsules each containing 1 tablet moxifloxacin.
  The participants received 2 tablets and 2 capsules at each dosing with approximately 150 ml water.
  Interventions: Drug: Placebo matching CG5503 PR tablet; Drug: Placebo matching moxifloxacin capsule; Drug: 400 mg Moxifloxacin tablet (overencapsulated)

INTERVENTIONS:
Drug: 100 mg CG5503 (tapentadol hydrochloride) PR tablet — 100 mg CG5503 (tapentadol hydrochloride) PR tablet.
  Arms: CG5503 PR 100 mg twice daily (tapentadol hydrochloride); CG5503 PR 200 mg twice daily (tapentadol hydrochloride)
Drug: Placebo matching CG5503 PR tablet — Matching placebo tablet to CG5503 PR tablet.
  Arms: CG5503 PR 100 mg twice daily (tapentadol hydrochloride); Moxifloxacin 800 mg single dose; Placebo
Drug: Placebo matching moxifloxacin capsule — Matching placebo capsule to moxifloxacin capsule.
Drug: 400 mg Moxifloxacin tablet (overencapsulated) — Overencapsulated 400 mg Moxifloxacin tablet.
  Arms: Moxifloxacin 800 mg single dose

SUMMARY:
The effect of multiple oral administration of two doses of CG5503 PR (prolonged release) compared to placebo on the electrical activity of the heart were investigated. The rationale to perform this study was to exclude any effect of CG5503 on the heart rhythm. This study was a randomised, double-blind, double-dummy, placebo- and moxifloxacin-controlled, 4-way cross-over study. Participants were given a combination of either CG5503 PR and placebo (medication with inactive ingredients which looks like the study drug) or moxifloxacin and placebo. Moxifloxacin was used as a positive control. It has consistently shown that it has an effect on the heart rhythm.

Within 14 days prior to the first dosing, participants had a physical examination, a 12-lead electrocardiogram (ECG) was recorded and haematological, serological, biochemical, and urine analyses took place. A blood sample for optional genotyping of genes responsible for long QT syndrome was taken. During each dosing session, the participants were confined in the evening before baseline assessments were performed and stayed in the clinic until 48 hours after the last dosing. Study medication was administered on Day 1 and 2 in the morning (0.5 hours after breakfast) and in the evening (1.5 hours after dinner), and on Day 3 in the morning (0.5 hours after breakfast). Dosing was separated by at least 7 days between the last dosing of each period and the first dosing of next period. Interim analysis of ECG-data were performed after completion of 24 participants (group 1) with possible subsequent adjustment of sample size for group 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian participants aged 45-65 years;
* Body mass index (BMI) between 19 and 27 kilograms/square meter inclusive;
* Participants must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram , vital signs, and clinical laboratory parameters (serum/urine biochemistry, serology and haematology). Electrocardiogram (ECG) parameters and vitals signs must be in the ranges given in exclusion criteria 3-8 and 11-14, respectively) Minor deviations of laboratory values from the normal range may be accepted (except potassium and magnesium), if judged by the investigator to have no clinical relevance and if not considered to interfere with the study objectives.
* Negative human immunodeficiency virus (HIV) 1/2 -antibodies, hepatitis B surface (HBs)-antigen, hepatitis B core (HBc)-antibodies and hepatitis C virus (HCV)-antibodies at the prestudy medical examination;
* Negative blood beta-human chorionic gonadotropine (HCG)-test for women of child bearing potential;
* Participants giving written consent to participate within this study;
* Participants giving written consent for blood sampling to be genotyped for genes responsible for long QT syndrome (KCNQ1, human ether-a-go-go-related gene (HERG), SCN5A, KCNE1, KCNE2, KCNJ2).

Exclusion Criteria:

* Regular use of any medication within four weeks prior to commencement of the study (self-medication or prescription except for hormonal contraception and HRT);
* Smoker more than 5 cigarettes per day;
* No regular sinus rhythm;
* ECG interval: QRS complex above 100 millisecond;
* ECG interval: PQ above 200 milliseconds;
* ECG interval: RR above 1333 milliseconds;
* QT/QTc intervals above 450 milliseconds;
* Known family history of sudden cardiac death and arrhythmias;
* Diseases and functional disorders of the gastrointestinal tract, liver, cardiovascular system or kidneys;
* Malignancy;
* History of orthostatic hypotension;
* Resting pulse rate below 45 beats/min or above 90 beats per minute;
* Systolic blood pressure above 160 mmHg or below 100 mmHg;
* Diastolic blood pressure above 95 mmHg or below 50 mmHg;
* History of drug allergy;
* Bronchial asthma;
* Participation in another clinical trial within the last three months before starting this study (exception: characterisation of metaboliser status);
* Blood donation (more than 100 milliliters) in the last three months before the start of the study;
* History or evidence of alcohol or drug abuse;
* Positive drug abuse screening test;
* Extremely unbalanced diet (in the opinion of the investigator);
* Excessive consumption of food or beverages containing caffeine (more than 1000 milliliters of coffee per day or other equivalent amounts of caffeine);
* Known or suspected of not being able to comply with the study protocol;
* Not able to communicate meaningfully with the investigator and staff;
* Neurotic personality, psychiatric illness, or suicide risk;
* History of seizures;
* Known hypersensitivity to opioids or quinolones;
* Pregnancy (for female participants);

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
The mean of corrected QT interval (QTc) differences on Day 3 at 3 to 7 hours to matched time points on Day 0 of the respective treatment period | Baseline (Day 0) to Day 3
  On Day 0 drug-free baseline 12-lead ECGs were recorded (in supine position after at least 10 minutes of rest) at time points corresponding to those on Day 3. On Day 3, 12-lead ECGs were recorded prior to and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 and 24 hours after dosing. A regression analysis was applied for each participant to obtain an individual correction.

SECONDARY OUTCOMES:
The differences of the QTc at each time point on Day 3 to the time matched QTc on Day 0 of each period | Baseline (Day 0) to Day 3
  In addition to the corrected QT by regression as described for the primary endpoint, QTc was calculated by the following formulas: Fridericia, Framingham, and Bazett.
Incidence of treatment emergent adverse events | Day 1 to Day 5
  Number of adverse events and number of participants with adverse events.
Withdrawal symptoms: 5 categories of COWS scale, sum of scores (of 11 items) and changes to placebo in sum of scores | Day 4 and Day 5
  The clinical opiate withdrawal scale (COWS) assessment consisted of 11 questions which rated the severity of opiate withdrawal symptoms, including resting pulse rate, gastrointestinal upset, sweating, restlessness, pupil size, tremor, anxiety or irritability, bone or joint aches, gooseflesh skin, yawning, and runny nose or tearing. Each symptom was rated on a scale from 0 (not present) to 4 or 5 (most severe). The total score was calculated by summing the 11 individual scores. Scores from 0 to 4 are considered "no withdrawal", from 5 to 12 "mild withdrawal", from 13 to 24 "moderate withdrawal", 25 to 36 "moderately severe withdrawal" and above 36 "severe withdrawal".
Pharmacokinetic parameter: Cmax(4-6h) of CG5503 base after the first dose | Day 1 to Day 5
  Maximum serum concentration in the observed time interval between 4 and 6 hours [Cmax(4-6h)]. Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration. Concentrations of CG5503 base in serum were determined by using validated High Performance Liquid Chromatography (HPLC) methods with fluorometric detection.
Pharmacokinetic parameter: tmax(4-6h) of CG5503 base after the first dose | Day 1 to Day 5
  Time to reach maximum serum concentration in the observed time interval between 4 and 6 hours [tmax(4-6h)]. Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: AUCss of CG5503 base after the last dose | Day 1 to Day 5
  Area under the concentration vs. time curve in dosing interval τ at steady state (AUCss). Blood samples for the determination of serum concentrations were taken at pre-dose and at up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: AUC of CG5503 base after the last dose | Day 1 to Day 5
  Area under the concentration vs. time curve (AUC) after the last dose. Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: AUCextr of CG5503 base after the last dose | Day 1 to Day 5
  Extrapolated part to infinity of AUC (AUCextr) after the last dose. Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: AUC%extr of CG5503 base after the last dose | Day 1 to Day 5
  Extrapolated part to infinity of AUC in percent (AUC%extr) after the last dose.
Pharmacokinetic parameter: Css,min of CG5503 base after the last dose | Day 1 to Day 5
  Minimum observed serum concentration during dosing interval τ at steady state (Css,min). Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: Css,max of CG5503 base after the last dose | Day 1 to Day 5
  Maximum observed serum concentration during dosing interval τ at steady state (Css,max). Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: Css,ave of CG5503 base after the last dose | Day 1 to Day 5
  Average serum concentration during dosing interval τ at steady state (Css,ave). Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: tss,max of CG5503 base after the last dose | Day 1 to Day 5
  Time to reach maximum serum concentration during dosing interval τ at steady state (tss,max). Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: λz of CG5503 base after the last dose | Day 1 to Day 5
  Apparent terminal elimination rate constant (λz) after the last dose. Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: t½,z of CG5503 base after the last dose | Day 1 to Day 5
  Apparent terminal half-life (t½,z) after the last dose. Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: CL/f of CG5503 base after the last dose | Day 1 to Day 5
  Apparent oral clearance at steady state (CL/f). Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: PTF (%) of CG5503 base after the last dose | Day 1 to Day 5
  Peak-trough fluctuation at steady state (PTF). Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.
Pharmacokinetic parameter: RA(Cmax) of CG5503 base after the last dose | Day 1 to Day 5
  Accumulation ratio (RA) calculated from Css,max at steady state and Cmax(4-6 hours) after single dosing. Blood samples for the determination of serum concentrations were taken at pre-dose and up to 12 hours on Day 1, prior to the morning and the evening dose on Day 2 and before and up to 48 hours after the last drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- DE001 - Contract research organisation, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No